CLINICAL TRIAL: NCT06283420
Title: Metabolic Response to the Initiation of Heart Failure Therapy (GliF Study)
Brief Title: Metabolic Response to the Initiation of Heart Failure Therapy
Acronym: GliF
Status: Recruiting | Type: Observational
Sponsor: Vojtech Melenovsky, MD, PhD (Other Government)
Responsible Party: Sponsor-Investigator, Vojtech Melenovsky, MD, PhD, Prof., Institute for Clinical and Experimental Medicine
Organization: Institute for Clinical and Experimental Medicine (Other Government)
Other Study IDs: CarDia_WP5_P1_IRB:25059/23
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure
Keywords: SGLT2 inhibitors; hypoxia; metabolism; HIF; sGC stimulators
MeSH Terms: conditions — Heart Failure; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma and DNA for analysis of genetic variants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HF patients initiated with sodium-glucose transport protein 2 (SGLT2) inhibitor: HF patients with medical indication to initiation of SGLT2 inhibitors
- HF patients initiated with soluble gluanylate cyclase (sGC) stimulator: HF patients with medical indication to initiation of sGC stimulator
- HF patients initiated with sacubitril/valsartan (ARNI): HF patients with medical indication to initiation of ARNI
- HF patients without change of their chronic medication: these HF patients (without ARNI, sGCs or SGLT2i) will serve as internal controls during observational part of the study (3 mo)

SUMMARY:
This protocol is a component of the CarDia project under the National Institute for Metabolic and Cardiovascular Disease Research (EXCELES Program, ID: LX22NPO5104), which is financed by the European Union - Next Generation EU. It falls under Work Package 5 (WP5), focusing on metabolic disorders in heart failure. The aim of this observational protocol is to track the biochemical and metabolomic reactions to the commencement of standard heart failure medications (SGLT2i, soluble guanylate cyclase-sGC stimulators, sacubitril/valsartan-ARNI) and to assess if the initial response (within the first three months) can predict the disease's progression. The protocol will investigate the temporal changes in parameters that indicate neurohumoral activation, hypoxia response, systemic energy substrate metabolism, iron metabolism, and HIF1A activation in peripheral blood following the initiation of standard heart failure therapy (baseline, 1 day, 1 week, 1 month, 3 months). This study could yield crucial insights into identifying individuals who exhibit a poorer response to the new treatment and are at a higher risk of an unfavorable disease trajectory. Patients will be compared with a control group, who are those without any therapy alteration during the initial observation period (3 months). As an observational study, the decision to initiate therapy will be based solely on medical indications. Heart failure patients at the Cardiocenter of the Institute for Clinical and Experimental Medicine - IKEM in Prague, CZ will undergo blood sampling at specific intervals before and after the initiation of clinically indicated treatment. A subset of patients will also receive genetic DNA testing to explore gene variability that influences the metabolic neurohumoral response to heart failure.

Patients will be followed up at 1 and 2-year intervals to monitor the occurrence of clinical events. The study's observational nature ensures that participation does not influence the standard of care or pharmacotherapy selection.

ELIGIBILITY:
Inclusion Criteria:

* ability to give written informed consent
* Heart failure New York Functional class (NYHA) II-IV with duration more than 3 months (regardless ejection fraction, universal definition of HF)
* NTproBNP more than 125 pg/ml at screening (Universal definition of HF)
* O2 sat more than 90%

Exclusion Criteria:

* Previous SGLT2 inhibitor therapy or i.v., iron therapy in past 3 months (for SGLT2i arm)
* Previous sGC stimulator (for sGC arm), or previous ARNI (for ARNI arm), or previous SGLT2i, sGC or ARNI for control group.
* Coronary artery bypass grafting (CABG), cardiac resynchronisation therapy (CRT), STEMI, valve replacement, in past 3 months, or planned within next 3 months
* Blood loss needing transfusion in past 3 months
* Clinical instability (including HF hospitalization) in the past 1 month
* Myelodysplasia, chronic hemolysis, erythropoetin therapy
* Systemic inflammatory condition (lupus, rheumatoid arthritis...) or infection
* Uncontrolled cancer
* Chronic kidney disease (CKD) grade 4-5
* Severe anemia with Hgb less than 90 g/L
* No chronic exposure to hypoxia (severe chronic obstructive pulmonary disease, obstructive sleep apnoea, long-term oxygen therapy)
* History of SGLT2i allergy or intolerance
* Repeated genitourinary infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable HF patients with HFrEF, HFmrEF or HFpEF
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
hematocrit | difference 3 mo-baseline
  full blood count hematocrit

SECONDARY OUTCOMES:
Hypoxia inducible factor (HIF) response | baseline, 1 day, 1 week, 1 mo and 3 mo after baseline
  gene expression of HIF1A-regulated genes in platelets
hepcidin | baseline, 3 months
  hepcidin plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical end Experimental Medicine - IKEM, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided